CLINICAL TRIAL: NCT02705326
Title: Evaluating the Efficacy of Opti-Speech, a 3D Visual Feedback System, for Speech Treatment
Brief Title: Evaluating the Efficacy of Opti-Speech for Speech Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vulintus, Inc. (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Callier Center for Communication Disorders (Unknown); Cleveland Hearing and Speech Center (Unknown); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VUL_2R44DC013467_OptiSpeech; 2R44DC013467 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-10 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-05

CONDITIONS: Articulation Disorder; Dysarthria; Prelingual Deafness
MeSH Terms: conditions — Articulation Disorders; Dysarthria; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Opti-Speech (Experimental): Speech treatment will be guided by Opti-Speech's visual feedback of tongue movement during speech
  Interventions: Device: Opti-Speech

INTERVENTIONS:
Device: Opti-Speech — Uses visual feedback of the tongue's motion to guide speech sound production

SUMMARY:
The purpose of this study is to determine if feedback from a three-dimensional real-time visualization of the tongue, a program called Opti-Speech, can be used to improve speech.

DETAILED DESCRIPTION:
Participants will be asked to complete the Goldman Fristoe Test of Articulation along with several other assessment tests. Then speech treatment, guided by Opti-Speech, will be provided to the participant for up to 10 treatment sessions. The participant will be asked to come back after the final treatment for a 2-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* English speaking individuals with speech errors resulting from persistent speech sound disorder, individuals with dysarthria resulting from neurological disorders and individuals with pre-lingual or congenital deafness.

Exclusion Criteria:

* Cognitive impairments that affect their ability to understand and follow instructions by the treating speech language pathologists

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Percent articulatory accuracy | within 30 minutes of treatment
  Sound probe lists will be administered within 30 minutes of treatment. Probe lists will be scored as correct or incorrect. The percentage of probes correct will be calculated

SECONDARY OUTCOMES:
Change in Accuracy of Speech Sound Production from Pre-Treatment to Post-Treatment | Immediately prior to first speech treatment and 2 months after final treatment.
  The Goldman Fristoe Test of Articulation will be administered prior to any speech treatment with Opti-Speech and again 2 months after the final speech treatment session. The percentage of consonants correct (PCC) will be used to assess the change in accuracy of speech sound production from pre-treatment to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jennell Vick, PhD, Principal Investigator — Cleveland Hearing and Speech Center, Case Western Reserve University; Thomas F Campbell, PhD, Principal Investigator — Callier Center for Communication Disorders at UT Dallas; Holle L Carey, MS, Principal Investigator — Vulintus, Inc.
Locations (2):
- United States (2):
  - The Cleveland Hearing and Speech Center, Cleveland, Ohio
  - Callier Center for Communication Disorders at UT Dallas, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Katz WF, Mehta S. Visual Feedback of Tongue Movement for Novel Speech Sound Learning. Front Hum Neurosci. 2015 Nov 19;9:612. doi: 10.3389/fnhum.2015.00612. eCollection 2015. PMID 26635571
- See also: Opti-Speech Demo — http://www.vulintus.com/optispeech/